CLINICAL TRIAL: NCT05594888
Title: GRIP: Evaluation of the Comparability of the Maximum Isometric Grip Strength Measurement Assessed With the JAMAR© Hydraulic Hand Dynamometer, the JAMAR© Smart Hand Dynamometer and the Martin Vigorimeter
Brief Title: GRIP: Maximum Isometric Grip Strength Assessed With Three Different Hand-held Dynamometers
Status: Completed | Type: Observational
Sponsor: Johannes Scherr (Other)
Responsible Party: Sponsor-Investigator, Johannes Scherr, Prof. Dr. med. Johannes Scherr, Balgrist University Hospital
Organization: Balgrist University Hospital (Other)
Other Study IDs: BASEC-Nr.:2022-01400
Record Dates: First submitted 2022-10-02; First posted 2022-10-26 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Grip
Keywords: Maximum isometric grip strength; Hand-held dynamometer; Reference values; Physical therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- PART 1- Group A: Male and female volunteers (age 18-64 years) working at University Hospital Balgrist. Assessment of validity and intrasubject reliability of maximum isometric grip strength assessed with:
  * JAMAR© Smart Dynamometer [kg]
  * JAMAR© Hydraulic Dynamometer [kg]
  * Martin Vigorimeter [kPa]
- PART 1 - Group B: Male and female volunteers (age 18-64 years) working at University Hospital Balgrist. Assessment of validity and intrasubject reliability and assessment of intersession reliability of maximum isometric grip strength assessed with:
  * JAMAR© Smart Dynamometer [kg]
  * JAMAR© Hydraulic Dynamometer [kg]
  * Martin Vigorimeter [kPa]
- PART 2: Male and female volunteers (age ≥ 10 years).
  Maximum isometric grip strength is assessed (no intervention):
  * JAMAR© Smart Dynamometer [kg]
  * JAMAR© Hydraulic Dynamometer [kg]
  * Martin Vigorimeter [KPa]

SUMMARY:
Maximum isometric grip strength (MIGS) is a cost-effective, easily accessible, valid and reliable outcome measure for assessing upper body strength in both, adults and children. The the JAMAR Hydraulic Hand Dynamometer is the current gold standard for measuring MIGS. For certain age- and activity-groups, alternative devices may be more appropriate. To date, the quality criteria (test-retest-reliability and validity) of the JAMAR Smart Hand Dynamometer and the Martin Vigorimeter compared to the current gold standard are not yet investigated. Furthermore, no reference values for different age-, sex-, or activity level groups exist with regard to underlying disease entities for these three devices.

DETAILED DESCRIPTION:
This quality analysis of test-retest reliability and validity (PART 1) serves as a basis for a further sensitivity analysis, whereby in a second step, a database with valid personalised age-, sex- and activity-related reference values for the respective measurement instrument, considering chronic concomitant diseases, is to be generated. The objectives of this study are therefore to 1) assess the test-retest reliability (intrasubject and intersession) and validity of JAMAR© Hydraulic and JAMAR© Smart dynamometers and Martin Vigorimeter (PART 1) and 2) undertake a sensitivity analysis providing valid personalised reference values for precision medicine (PART 2).

Thus, no study has yet comprehensively investigated all relevant influencing factors in a single and thus homogeneous study setting, so bias can be expected from this alone. The findings of this two-step study should enable physicians and therapists to compare the grip strength measurements of their patients with normative values in relation to their age, sex and activity group, as well as to any underlying chronic diseases that may be present. This allows realistic treatment and training goals to be set and patient performance to be interpreted.

ELIGIBILITY:
Inclusion Criteria Part 1:

* Male and female volunteers with age 18-64 years
* Body mass index < 30 kg/m2
* Informed consent signed

Inclusion Criteria Part 2:

* Male and female volunteers with age ≥ 10 years
* Informed consent signed (if age < 14 years, signed by parents or legal guardians)

Exclusion Criteria Part 1 and 2:

* Disease or injury (e.g., musculoskeletal or neurological) that could affect upper extremity strength
* Physical impairment of the upper extremity (visible swelling or the presence of a splint or cast)
* Acute pain or infection
* Cognitive impairment (inability to understand and/or follow directions)
* Insufficient language of the German language

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Part 1:
  * Male and female volunteers (age 18-64 years) working at University Hospital Balgrist.
  * 40 participants: to exclude possible sex aspects, ratio ♀: ♂ = 1:1
  Part 2:
  * Male and female volunteers (age ≥ 10 years). MIGS is used as a health indicator throughout different age- and sex groups.
  * 20 participants per age-group and sex with a total of 520 subjects are planned
Sampling Method: Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
PART 1: Quality criteria: Intrasubject reliability | 5 minutes
  Test-retest reliability of the JAMAR© Smart Dynamometer, the JAMAR© Hydraulic Dynamometer and Martin Vigorimeter measuring MIGS will be assessed by intrasubject realiability.
  --> 5 attempts per device and dominant/adominant hand will be measured.
PART 1: Quality criteria: Intersession reliability | 5 minutes
  Test-retest reliability of the JAMAR© Smart Dynamometer, the JAMAR© Hydraulic Dynamometer and Martin Vigorimeter measuring MIGS will be assessed by intersession realiability.
  --> 5 attempts per device and dominant/adominant hand at two different days will be measured.
PART 1: Quality criteria: Validity | 5 minutes
  Validity of the JAMAR© Smart Dynamometer, the JAMAR© Hydraulic Dynamometer and Martin Vigorimeter measuring MIGS will be assessed by plotting the differences in grip force measurements of the 3 measurement devices against their means, with ± 1.96 SD as cut-off values (limits of agreement).
  --> 5 attempts per device and dominant/adominant hand will be measured.
PART 2: Comparability of MIGS measurement | 10 minutes
  Evaluation of comparability of MIGS measurement assessed with the JAMAR© Smart Dynamometer, the JAMAR© Hydraulic Dynamometer and the Martin Vigorimeter
  -> Best out of 3 attempts per device and dominant/adominant hand

SECONDARY OUTCOMES:
PART 2: Age-specific refence values - JAMAR© Hydraulic | 1 minute
  Age-specific refence values for MIGS assessed with the JAMAR© Hydraulic. Age is assessed by the number of years. Thirteen age groups are established with an increment of five to ten years: 10-14/15-19/20- 29/30-39/40-44/45-49/50-54/55-59/60-64/65-69/70-74/75-79/80+
PART 2: Age-specific refence values - JAMAR© Smart | 1 minute
  Age-specific refence values for MIGS assessed with the JAMAR© Smart. Age is assessed by the number of years. Thirteen age groups are established with an increment of five to ten years: 10-14/15-19/20- 29/30-39/40-44/45-49/50-54/55-59/60-64/65-69/70-74/75-79/80+
PART 2: Age-specific refence values - Martin Vigorimeter | 1 minute
  Age-specific refence values for MIGS assessed with the Martin Vigorimeter. Age is assessed by the number of years. Thirteen age groups are established with an increment of five to ten years: 10-14/15-19/20- 29/30-39/40-44/45-49/50-54/55-59/60-64/65-69/70-74/75-79/80+
PART 2: Sex-specific refence values - JAMAR© Hydraulic | 0.5 minute
  Sex-specific refence values for MIGS assessed with the , JAMAR© Hydraulic. Sex is recorded as male or female (biological sex).
PART 2: Sex-specific refence values - JAMAR© Smart | 0.5 minute
  Sex-specific refence values for MIGS assessed with the JAMAR© Smart. Sex is recorded as male or female (biological sex).
PART 2: Sex-specific refence values - Martin Vigorimeter | 0.5 minute
  Sex-specific refence values for MIGS assessed with the Martin Vigorimeter. Sex is recorded as male or female (biological sex).
PART 2: Physical activity-specific reference values - JAMAR© Hydraulic | 2 minutes
  Physical activity-specific reference values for MIGS measurements assessed with the JAMAR© Hydraulic.
  The IPAQ, the PAQ-A and the PAQ-C are used to assess individual levels of physical activity through all age groups. The IPAQ is a reliable and valid instrument that shows very good repeatability, was designed for people aged 18-65 years and is validated for persons aged 18-84 years. Adolescents between 15 and 18 years of age are assessed using the PAQ-A and children aged 10-14 years are assessed by the PAQ-C.
PART 2: Physical activity-specific reference values - JAMAR© Smart | 2 minutes
  Physical activity-specific reference values for MIGS measurements assessed with the JAMAR© Smart.
  The IPAQ, the PAQ-A and the PAQ-C are used to assess individual levels of physical activity through all age groups. The IPAQ is a reliable and valid instrument that shows very good repeatability, was designed for people aged 18-65 years and is validated for persons aged 18-84 years. Adolescents between 15 and 18 years of age are assessed using the PAQ-A and children aged 10-14 years are assessed by the PAQ-C.
PART 2: Physical activity-specific reference values - Martin Vigorimeter | 2 minutes
  Physical activity-specific reference values for MIGS measurements assessed with the Martin Vigorimeter.
  The IPAQ, the PAQ-A and the PAQ-C are used to assess individual levels of physical activity through all age groups. The IPAQ is a reliable and valid instrument that shows very good repeatability, was designed for people aged 18-65 years and is validated for persons aged 18-84 years. Adolescents between 15 and 18 years of age are assessed using the PAQ-A and children aged 10-14 years are assessed by the PAQ-C.
PART 2: Refence values for subjects with different disease entities - JAMAR© Hydraulic | 1 minute
  Refence values for subjects with different disease entities that might influence target value of MIGS measurement assessed with the JAMAR© Hydraulic
  Any chronic disease entities that may be present, (possible chronic diseases according to organ class) are recorded:
  * Pulmonary (e.g., COPD)
  * Cardiac (e.g., CHF)
  * Neurological (apoplexy, PNP)
  * Gastroenterological (e.g., chronic gastritis)
  * Gynaecological (e.g., endometriosis)
  * Rheumatic (e.g., arthritis)
  * Oncological
  * Musculoskeletal (e.g., spine, lower extremities)
  * Metabolic (e.g., diabetes mellitus).
PART 2: Refence values for subjects with different disease entities - JAMAR© Smart | 1 minute
  Refence values for subjects with different disease entities that might influence target value of MIGS measurement assessed with the JAMAR© Smart
  Any chronic disease entities that may be present, (possible chronic diseases according to organ class) are recorded:
  * Pulmonary (e.g., COPD)
  * Cardiac (e.g., CHF)
  * Neurological (apoplexy, PNP)
  * Gastroenterological (e.g., chronic gastritis)
  * Gynaecological (e.g., endometriosis)
  * Rheumatic (e.g., arthritis)
  * Oncological
  * Musculoskeletal (e.g., spine, lower extremities)
  * Metabolic (e.g., diabetes mellitus).
PART 2: Refence values for subjects with different disease entities - Martin Vigorimeter. | 1 minute
  Refence values for subjects with different disease entities that might influence target value of MIGS measurement assessed with the Martin Vigorimeter.
  Any chronic disease entities that may be present, (possible chronic diseases according to organ class) are recorded:
  * Pulmonary (e.g., COPD)
  * Cardiac (e.g., CHF)
  * Neurological (apoplexy, PNP)
  * Gastroenterological (e.g., chronic gastritis)
  * Gynaecological (e.g., endometriosis)
  * Rheumatic (e.g., arthritis)
  * Oncological
  * Musculoskeletal (e.g., spine, lower extremities)
  * Metabolic (e.g., diabetes mellitus).
PART 1 + 2: General health | 10 minutes
  The OSTRC questionnaire is used to assess general health before the first study appointment.
  The OSTRC contains four key questions recording the level of participation and performance impairment and the degree of symptoms caused by injury or illness. A severity score is then calculated based on these four questions.

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Scherr, Prof Dr med, Principal Investigator — Balgrist University Hospital
Locations (1):
- University Hospital Balgrist, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided